CLINICAL TRIAL: NCT01161667
Title: A Single Dose, Two-Period, Two-Treatment, Two-Way Crossover Bioequivalence Study of Naratriptan Hydrochloride 2.5 mg Tablets Under Fasted Conditions
Brief Title: Bioequivalency Study of Naratriptan Hydrochloride 2.5 mg Under Fasted Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roxane Laboratories (Industry)
Responsible Party: Elizabeth Ernst, Cirector, Drug Regulatory and Medical Affairs, Roxane Laboratories, Inc.
Organization: West-Ward Pharmaceutical (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NARA-T25-PVFS-1
Record Dates: First submitted 2010-07-12; First posted 2010-07-13 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — naratriptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: naratriptan hydrochloride — 2.5 mg tablet
  Other Names: AMERGE

SUMMARY:
The objective of this study was to prove the bioequivalence of Naratriptan Hydrochloride Tablet under fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal findings on the physical examination, medical history, or clinical laboratory results during screening

Exclusion Criteria:

* Positive test for HIV, Hepatitis B, or Hepatitis C.
* Treatment with known enzyme altering drugs.
* History of allergic or adverse response to naratriptan hydrochloride or any comparable or similar product.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2007-09; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
bioequivalence determined by statistical comparison Cmax | 9 days

CONTACTS AND LOCATIONS:
Overall Officials: Linda Bavisotto, M.D., Principal Investigator — Charles River Northwest Kinetics
Locations (1):
- Charles River Northwest Kinetics, Tacoma, Washington, United States